CLINICAL TRIAL: NCT00290173
Title: Ritodrine in Oral Maintenance of Tocolysis After Active Preterm Labor: Randomized Controlled Trial
Brief Title: Ritodrine in Oral Maintenance of Tocolysis After Active Preterm Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zagreb (Other)
Collaborators: Ministry of Science, Education and Sport, Republic of Croatia (Other Government)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0129111
Record Dates: First submitted 2006-02-08; First posted 2006-02-10 (Estimated); Last update posted 2006-05-04 (Estimated); Status verified 2006-02

CONDITIONS: Pregnancy
Keywords: pre term labor; therapy; maintenance

INTERVENTIONS:
Drug: efficacy of oral ritodrine in maintaining uterine quiescence

SUMMARY:
This is a trial comparing the efficacy of oral ritodrine in the form of sustained release capsules for the maintenance of uterine quiescence after successfully treated episode of threatened preterm labor.

DETAILED DESCRIPTION:
We randomized 120 women with singleton pregnancy who were successfully treated for threatened preterm labor before 34 completed weeks to receive either maintenance tocolysis with two 40 mg ritodrine sustained release capsules three times a day (study group, n=62) or no treatment (control group, n=58) for three days. The primary outcome measure was the recurrent episode of threatened preterm labor within 72 hours, which was defined as regular palpable uterine contractions and change in cervical effacement and/or cervical dilatation on clinical examination. Secondary outcome measures included the incidence of preterm birth, neonatal adverse outcomes, and maternal side effects.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy between completed 24 to 24 weeks
* Successfully treated episode of threatened preterm labour by intravenous preparations
* No uterine contractions

Exclusion Criteria:

* Uterine contractions (painful, clinically palpable, or present on cardiotocography)
* Cervical dilatation of ≥5 cm
* Clinical and laboratory signs of infection defined as offensive vaginal discharge on clinical examination, vaginal pH ≥5, white blood cell (WBC) count >16×109/L, and C-reactive protein (CRP) >10 mg/L
* Positive findings of microorganisms rather than normal vaginal flora on high vaginal swab
* Any signs of fetal distress according to cardiotocography, Doppler assessment of blood flow in umbilical artery, and biophysical profile of <8.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Study Completion 2005-08

PRIMARY OUTCOMES:
the recurrence of preterm labor within 72 hours after discontinuation of IV treatment

SECONDARY OUTCOMES:
Secondary outcome measures were incidence of preterm delivery before 37 weeks of gestation, incidence of early preterm delivery before completed 34 weeks of gestation, prolongation of pregnancy, birth weight, perinatal mortality and perinatal morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Ozren Grgic, MD, Principal Investigator — Sveti Duh Hospital; Ratko Matijevic, MD,PhD, Study Chair — Sveti Duh Hospital
Locations (1):
- Department of Obstetrics and Gynecology, University of Zagreb, Zagreb, Croatia

REFERENCES:
- [Result] Matijevic R, Grgic O, Vasilj O. Ritodrine in oral maintenance of tocolysis after active preterm labor: randomized controlled trial. Croat Med J. 2006 Feb;47(1):25-31. PMID 16489694